CLINICAL TRIAL: NCT06488027
Title: DAO DEFICIENCY SCREENING AMONG PATIENTS WITH INSOMNIA SYMPTOMS
Status: Completed | Type: Observational
Sponsor: AB Biotek (Industry)
Responsible Party: Sponsor
Other Study IDs: DAO-SLEEP-2022
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Insomnia; Insomnia Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with insomnia symptoms: Patients with insomnia symptoms visiting AdSalutem sleep center

SUMMARY:
Insomnia is prevalent in the global population. Diamino oxidase (DAO) is an enzyme that degrades histamine. When there is not enough DAO enzyme activity in the body, histamine accumulates and it can lead to symptoms in the nervous system, among others. In this study we wanted to study the prevalence of DAO deficiency in pacients with insomnia symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old
* With one or more symptoms of insomnia
* Explicit acceptance to participate to the study through informed consent

Exclusion Criteria:

* Insomnia symptoms that could be justified by the existance of another sleep pathology (e.g., narcolepsy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with insomnia symptoms attending AdSalutem sleep center
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
number of patients with insomnia symptoms and DAO deficiency | at the time of enrollment
  number (absolute and percentage) of patients with insomnia symptoms and DAO deficiency

CONTACTS AND LOCATIONS:
Overall Officials: Julia Ferrer Garcia, MSc, Study Chair — AdSalutem Sleep Institute
Locations (1):
- AdSalutem Sleep Institute, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Antropometric data
Supporting Information: Study Protocol, ICF, CSR
Time Frame: According to legislation
URL: https://www.abbiotekhealth.com/en/about-us/

REFERENCES:
- [Background] Schnedl WJ, Lackner S, Enko D, Schenk M, Holasek SJ, Mangge H. Evaluation of symptoms and symptom combinations in histamine intolerance. Intest Res. 2019 Jul;17(3):427-433. doi: 10.5217/ir.2018.00152. Epub 2019 Mar 7. PMID 30836736
- [Background] Garcia-Martin E, Ayuso P, Martinez C, Agundez JA. Improved analytical sensitivity reveals the occurrence of gender-related variability in diamine oxidase enzyme activity in healthy individuals. Clin Biochem. 2007 Nov;40(16-17):1339-41. doi: 10.1016/j.clinbiochem.2007.07.019. Epub 2007 Aug 11. PMID 17826755
- [Background] Ayuso P, Garcia-Martin E, Martinez C, Agundez JA. Genetic variability of human diamine oxidase: occurrence of three nonsynonymous polymorphisms and study of their effect on serum enzyme activity. Pharmacogenet Genomics. 2007 Sep;17(9):687-93. doi: 10.1097/FPC.0b013e328012b8e4. PMID 17700358
- [Derived] Lopez Garcia R, Ferrer-Garcia J, Sansalvador A, Quera-Salva MA. Prevalence of Diamine Oxidase Enzyme (DAO) Deficiency in Subjects with Insomnia-Related Symptoms. J Clin Med. 2024 Aug 6;13(16):4583. doi: 10.3390/jcm13164583. PMID 39200725